CLINICAL TRIAL: NCT06649435
Title: Seerlinq: a Non-invasive System for Remote Monitoring of Left Ventricular Filling Pressure in Heart Failure Patients
Brief Title: Seerlinq: Non-invasive LVFP Monitoring in HF
Acronym: PPG-HF
Status: Completed | Type: Observational
Sponsor: Seerlinq s. r. o. (Other)
Collaborators: Premedix Academy (Other)
Responsible Party: Sponsor
Other Study IDs: 2023001
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Photoplethysmography; Right Heart Catheterization
Keywords: heart failure; photoplethysmography; right heart catheterization
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- RHC cohort: Patients undergoing right heart catheterization (RHC) for invasive measurement of LVFP.
  Interventions: Procedure: PPG measurement
- ECHO cohort: Patients in whom LVFP (normal vs. elevated) will be classified non-invasively using transthoracic echocardiography (TTE).
  Interventions: Procedure: PPG measurement
- RPM cohort: Patients participating in a pilot remote patient monitoring program with regular home-based measurements.

INTERVENTIONS:
Procedure: PPG measurement — PPG signal will be measured on CE certified medical devices. Two measurements will be performed - standing and in the recumbent position using reflectance and transmitance method on finger and in ear canal. The each measurement will be 120s long.
  Detailed analysis of PPG signal and pathophysiological phenomena associated with HF - peripheral volume changes detectable in PPG signal - will help to understand better and clarify the pathophysiological mechanisms of peripheral volume changes in a failing heart.
  Groups: ECHO cohort; RHC cohort

SUMMARY:
Left ventricular filling pressure (LVFP) monitoring has been associated with improved quality of life, survival and reduced hospitalization rates. However, current LVFP monitoring methods are invasive, costly, and require long-term antithrombotic therapy.

The purpose of this study is to validate Seerlinq HeartCore, a novel CE-certified, non-invasive system that enables remote LVFP monitoring using photoplethysmography (PPG) and machine learning-based signal analysis.

DETAILED DESCRIPTION:
Heart failure (HF) affects approximately 1-2% of the adult population in developed countries, with prevalence exceeding 10% among individuals older than 70 years. Despite advancements in diagnostics and treatment guided by evidence-based medicine, HF remains associated with high morbidity and mortality; up to 17% of patients die and up to 44% require hospitalization within 12 months.

Monitoring of left ventricular filling pressure (LVFP) has been shown to improve survival, quality of life, and reduce hospitalization rates in patients with HF. However, existing methods for LVFP assessment are invasive, costly, and require long-term antithrombotic therapy, limiting their widespread application.

The purpose of this study is to validate HeartCore, a novel CE-certified, non-invasive system that enables remote LVFP monitoring using photoplethysmography (PPG) combined with machine learning-based signal analysis.

This will be a prospective, multicenter study enrolling three patient cohorts:

RHC cohort, ECHO cohort, and RPM cohort. Participants will undergo 120-second PPG recordings in both upright and supine positions using a standard pulse oximeter connected to a smartphone. The PPG signals will be transmitted to a secure server and processed by the HeartCore algorithm to estimate LVFP, expressed as the diastolic reserve index (DRI), where a higher DRI indicates lower LVFP.

The primary outcomes of the study will be:

* The discrimination performance of the PPG-based HeartCore system for detecting elevated LVFP in the RHC and ECHO cohorts, measured by receiver operating characteristic area under the curve (ROC AUC), sensitivity, and specificity.
* The change in DRI following furosemide up-titration in the RPM cohort.

The secondary outcome will be:

• The correlation between DRI and pulmonary capillary wedge pressure (PCWP) in the RHC cohort.

This study aims to demonstrate that a non-invasive, widely available, and scalable PPG-based system can provide reliable assessment of LVFP in HF patients, potentially improving the management and outcomes of this population.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged ≥ 18 years
* Able to understand, and willing to provide written ICF
* Stated willingness to comply with all study procedures
* Confirmed diagnosis of heart failure according to the 2021 ESC guidelines

Exclusion Criteria:

* Pregnancy or female participant lactating
* Advanced renal failure (glomerular filtration rate <25 ml/min or need for renal replacement therapy),
* Active malignancy requiring chemotherapy or radiotherapy
* Complex congenital heart disease
* Ventricular assist device support
* Pulmonary hypertension classified as WHO group 1 or groups 3-5.
* Other possible unforeseen medical conditions that the investigator deems unsafe for study participation

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 131 adult participants aged ≥ 18 years with diagnosed HF, enrolled into three cohorts - RHC, ECHO, RPM, fulfilling all the inclusion and none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Discrimination performance for elevated LVFP, measured by ROC AUC, sensitivity, and specificity in the ECHO studies. | in 1 year
  The ability to distinguish elevated left ventricular filling pressure (LVFP) will be assessed using receiver operating characteristic area under the curve (ROC AUC), sensitivity, and specificity metrics in echocardiogram (ECHO) studies. This evaluation aims to validate the diagnostic accuracy of the proposed method.
Discrimination performance for elevated LVFP, measured by ROC AUC, sensitivity, and specificity in the RHC studies. | in 1 year
  The ability to distinguish elevated left ventricular filling pressure (LVFP) will be assessed using receiver operating characteristic area under the curve (ROC AUC), sensitivity, and specificity metrics in right heart catheterization (RHC) studies. This evaluation aims to validate the diagnostic accuracy of the proposed method.
LVFP changes post-diuretic up-titration in the remote monitoring analysis, evaluating its role in monitoring treatment response. | in 1 year
  Changes in left ventricular filling pressure (LVFP) following diuretic up-titration will be analyzed through remote monitoring to assess its effectiveness in tracking treatment response. The change in LVFP (DRI) pre- and post-treatment adjustment will be compared using appropriate statistical method. This endpoint will explore the utility of continuous monitoring in optimizing heart failure management.

SECONDARY OUTCOMES:
The correlation between LVFP determined by PPG analysis by the Seerlinq HeartCore and LVFP (PCWP) measured during RHC. | in 1 year
  The correlation between left ventricular filling pressure (LVFP) estimated via photoplethysmography (PPG) analysis using the Seerlinq HeartCore device and LVFP (pulmonary capillary wedge pressure, PCWP) measured during right heart catheterization (RHC) will be evaluated. This correlation will help validate the PPG-based method as a non-invasive alternative for LVFP assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Böhm, MD, Principal Investigator — Seerlinq
Locations (1):
- Seerlinq s.r.o., Bratislava, Nové Mesto, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ponikowski P, Voors AA, Anker SD, Bueno H, Cleland JGF, Coats AJS, Falk V, Gonzalez-Juanatey JR, Harjola VP, Jankowska EA, Jessup M, Linde C, Nihoyannopoulos P, Parissis JT, Pieske B, Riley JP, Rosano GMC, Ruilope LM, Ruschitzka F, Rutten FH, van der Meer P; ESC Scientific Document Group. 2016 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: The Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC)Developed with the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2016 Jul 14;37(27):2129-2200. doi: 10.1093/eurheartj/ehw128. Epub 2016 May 20. No abstract available. PMID 27206819
- [Background] Crespo-Leiro MG, Metra M, Lund LH, Milicic D, Costanzo MR, Filippatos G, Gustafsson F, Tsui S, Barge-Caballero E, De Jonge N, Frigerio M, Hamdan R, Hasin T, Hulsmann M, Nalbantgil S, Potena L, Bauersachs J, Gkouziouta A, Ruhparwar A, Ristic AD, Straburzynska-Migaj E, McDonagh T, Seferovic P, Ruschitzka F. Advanced heart failure: a position statement of the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2018 Nov;20(11):1505-1535. doi: 10.1002/ejhf.1236. Epub 2018 Jul 17. PMID 29806100
- [Background] Silber HA, Trost JC, Johnston PV, Maughan WL, Wang NY, Kasper EK, Aversano TR, Bush DE. Finger photoplethysmography during the Valsalva maneuver reflects left ventricular filling pressure. Am J Physiol Heart Circ Physiol. 2012 May 15;302(10):H2043-7. doi: 10.1152/ajpheart.00609.2011. Epub 2012 Mar 2. PMID 22389389